CLINICAL TRIAL: NCT00776971
Title: Carbonated Soft Drinks May Alter Appetite Sensation and Appetite-Regulating Hormone Level and Lead to Increased Energy Intake.
Brief Title: Effect of Carbonated Soft Drinks on Appetite-Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: LG Life Sciences (Industry)
Responsible Party: Bjørn Richelsen/ Professor, Aarhus University Hospital
Model: Crossover | Masking: None
Other Study IDs: 20070134A
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2008-10-22 (Estimated); Status verified 2008-08

CONDITIONS: Obesity; Diet
MeSH Terms: conditions — Obesity | interventions — Sugar-Sweetened Beverages; Diet, Fat-Restricted; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sugar-sweetened soft drink (Experimental): 54g sugar/L, 180kJ/100mL
  Interventions: Other: Sugar-sweetened soft drink
- Aspartame-sweetened soft drink (Experimental): 1.5kJ/100mL
  Interventions: Other: Aspartame-sweetened soft drink
- Semi-skimmed milk (Active Comparator): 202kJ/100mL
  Interventions: Other: Semi-skimmed milk
- Water (Placebo Comparator): 0kJ/100mL
  Interventions: Other: Water

INTERVENTIONS:
Other: Sugar-sweetened soft drink — 500mL as a preload drink
  Arms: Sugar-sweetened soft drink
Other: Aspartame-sweetened soft drink — 500mL as a preload drink
  Arms: Aspartame-sweetened soft drink
Other: Semi-skimmed milk — 500mL as a preload drink
  Arms: Semi-skimmed milk
Other: Water — 500mL as a preload drink
  Arms: Water

SUMMARY:
Compared to solid foods, the nutritional energy of drinks may bypass the appetite regulation leading to obesity development. Although drinks sweetened with aspartame are available the anticipated positive effect of these drinks on obesity development has not been convincing. However, the mechanisms linking drinks intake to obesity are yet to be clarified.

The investigators aim is to investigate the short-term effects of soft drinks (sugar-sweetened and artificially sweetened (aspartame)), milk and water on the concentration of circulating appetite-regulating hormones, the subjective sensations of hunger and satiety (measured by visual analogue scales) and energy intake. The study is a crossover, intervention trial with 24 overweight, healthy volunteers. The subjects will be tested on four separate days for four hours. Each test day a preload drink (sugar-sweetened soft drink, aspartame-sweetened soft drink, semi-skimmed milk or water) is served.

The investigators expect to clarify the mechanisms linking drinking habits to obesity development and provide scientifically based nutritional guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-50 years;
* BMI between 28-36 kg/m2;
* Weight stabile 3 months prior to the study inclusion;
* Less than 10 hours of weekly exercise.

Exclusion Criteria:

* Diabetes
* Allergic to phenylalanine or milk
* Smoking
* Pregnancy or breast-feeding

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Four hours

SECONDARY OUTCOMES:
Appetite-regulating hormones, Glucose, Insulin; Energy intake | Four hours

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Richelsen, Professor, Study Chair — Department of Internal Medicine/Endocrinology C, Aarhus University Hospital
Locations (1):
- Department of Internal Medicine/Endocrinology C, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Maersk M, Belza A, Holst JJ, Fenger-Gron M, Pedersen SB, Astrup A, Richelsen B. Satiety scores and satiety hormone response after sucrose-sweetened soft drink compared with isocaloric semi-skimmed milk and with non-caloric soft drink: a controlled trial. Eur J Clin Nutr. 2012 Apr;66(4):523-9. doi: 10.1038/ejcn.2011.223. Epub 2012 Jan 18. PMID 22252107